CLINICAL TRIAL: NCT00047580
Title: A Multicenter, Open-Label, Randomized, 4-Way Crossover Trial of the Safety and Efficacy of Tizanidine Hydrochloride Capsules Versus Zanaflex (Tizanidine Hydrochloride) Tablets Taken Under Fed and Fasted Conditions in Patients With Moderate to Severe Spasticity
Brief Title: Comparison of Safety and Efficacy of Tizanidine Hydrochloride Capsules Versus Zanaflex® (Tizanidine Hydrochloride Tablets) Taken While in the Fed State (Just After a Meal) and in the Fasted State (Before a Meal) in Patients With Moderate to Severe Spasticity.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Elan Pharmaceuticals (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ELN021-502
Record Dates: First submitted 2002-10-08; First posted 2002-10-10 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis; Muscle Spasticity; Spinal Cord Injury; Stroke
Keywords: Spasticity; spasticity secondary to Multiple Sclerosis; Spinal Cord Injury; Stroke
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity; Spinal Cord Injuries; Stroke | interventions — tizanidine

INTERVENTIONS:
Drug: tizanidine hydrochloride capsule

SUMMARY:
This study is being conducted to compare the impact of somnolence (sleepiness) on cognition (awareness) as well as the safety and effectiveness of tizanidine hydrochloride capsules versus Zanaflex® (tizanidine hydrochloride tablets) taken while in the fed state (just after a meal) and in the fasted state (before a meal) in patients with moderate to severe spasticity.

ELIGIBILITY:
Inclusion Criteria:

* IRB approved ICF must be signed and dated by patient or patient's legal representative
* Male or Female 18 years of age or older
* Clinical diagnosis of established spasticity (at least 3 months) secondary to multiple sclerosis, stroke, or spinal cord injury
* Currently on stable dose of up to 36mg of Zanaflex
* Must be able to swallow tablets or capsules whole

Exclusion Criteria:

* Patients with dementia, aphasia, or other deficits in cognition
* Unwilling or unable to complete cognition test or daily diary
* Known sensitivity to Zanaflex
* Taking Zanaflex on an as needed ("prn") basis
* Currently being treated with drugs having significant effects at the alpha2 receptors whether agonist (i.e., clonidine, methyldopa) or antagonist (i.e., phenothiazines, imipramine)
* Currently on any other muscle relaxant or any drugs having muscle relaxant properties (including baclofen, dantrolene, diazepam and other benzodiazepines, tranquilizers, narcotic analgesics, high dose neuroleptics, chlormezanone, meprobamate, methocarbamol, orphenadrine, carisoprodol, gabapentin and clonidine
* Taking any over-the-counter or prescription sleep aids within 30 days prior to screening
* Use of illegal drugs or legal drugs for recreational purposes or excessive use of alcohol
* Patients suffering from disabling, symptomatic hypotension (i.e., syncope)
* Patients having any systemic disease such as renal insufficiency, clinically relevant elevations in hepatic transaminase, severe, uncontrolled systemic hypertension
* Any clinically significant illnesses, within four weeks of screening
* Patients with known sleep disorders
* Patients who participated in a clinical trial within thiry days prior to screening
* Women of childbearing potential who are pregnant, have a positive serum pregnancy test, lactating, or do not or will not take adequate contraceptive precautions for the duration of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2002-06; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Radiant Research, Tucson, Arizona
  - The Neurology Center, Encinitas, California
  - Northridge Neurological Center, Northridge, California
  - The Neurology Center, Oceanside, California
  - Neurology Medical Group of Diablo Valley, Walnut Creek, California
  - Colorado Neurology Movement Disorders Center, Englewood, Colorado
  - Yale Center for MS Treatment and Research, New Haven, Connecticut
  - Neurology Clinic Research Institution, Plantation, Florida
  - Axiom Clinical Research, Tampa, Florida
  - Comprehensive Neurology Specialists, PC, Atlanta, Georgia
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Springfield Clinic Neuroscience Institute, Springfield, Illinois
  - The Minneapolis Clinic of Neurology, Ltd., Minneapolis, Minnesota
  - Neurological Associates of Tulsa, Inc., Tulsa, Oklahoma
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - Sargent Rehabilitation Center, Warwick, Rhode Island